CLINICAL TRIAL: NCT03921411
Title: A Multicenter, Open-Label, Single-Group Clinical Trial to Assess the Pharmacokinetics and Safety of Nemolizumab (CD14152) in Adolescent Subjects (12-17 Years) With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Pharmacokinetics and Safety Study of Nemolizumab in Adolescent Participants With Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.116912
Record Dates: First submitted 2019-03-29; First posted 2019-04-19 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
Keywords: Nemolizumab; Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nemolizumab (Experimental): Nemolizumab
  Interventions: Biological: Nemolizumab

INTERVENTIONS:
Biological: Nemolizumab — Participants received subcutaneous (SC) injection of 30 milligram (mg) of Nemolizumab every 4 weeks (Q4W) over a 16-week treatment period, with a loading dose of 60 mg on Day 1.

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics and safety of nemolizumab in adolescent participants with AD.

ELIGIBILITY:
Key Inclusion Criteria

* Male or female participants ≥ 12 to < 17 years of age
* Chronic AD that has been documented for at least 2 years
* Eczema Area and Severity Index (EASI) score ≥ 16
* Investigator's Global Assessment (IGA) score ≥ 3
* AD involvement ≥ 10% of Body Surface Area (BSA)
* Documented recent history of inadequate response to topical medications
* Women of childbearing potential must agree to be strictly abstinent or to use an effective and approved method of contraception throughout the study and for 12 weeks after the last study drug injection.

Key Exclusion Criteria

* Body weight < 30 kilogram (kg)
* Cutaneous infection within 1 week or any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics, or antifungals within 1 week
* History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, example., monoclonal antibody)
* Any medical or psychological condition, or any clinically relevant laboratory abnormalities that may have put the subject at significant risk according to the investigator's judgment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Galderma Investigational Site, Fountain Valley, California
  - Galderma Investigational Site, Fremont, California
  - Galderma Investigational Site, Jacksonville, Florida
  - Galderma Investigational Site, Tampa, Florida
  - Galderma Investigational Site, Columbus, Georgia
  - Galderma Investigational Site, Sandy Springs, Georgia
  - Galderma Investigational Site, Gresham, Oregon
  - Galderma Investigational Site, Dallas, Texas
  - Galderma Investigational Site, Frisco, Texas
  - Galderma Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sidbury R, Alpizar S, Laquer V, Dhawan S, Abramovits W, Loprete L, Krishnaswamy JK, Ahmad F, Jabbar-Lopez Z, Piketty C. Pharmacokinetics, Safety, Efficacy, and Biomarker Profiles During Nemolizumab Treatment of Atopic Dermatitis in Adolescents. Dermatol Ther (Heidelb). 2022 Mar;12(3):631-642. doi: 10.1007/s13555-021-00678-7. Epub 2022 Jan 28. PMID 35088348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 participants were screened, of which 20 were enrolled and 18 participants were treated with study drug.
Period: Overall Study
Arm/Group | Nemolizumab
Started | 20
Treated | 18
Completed | 15
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Deviation | 2
Not completed — Enrolled, but never treated | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants who signed informed consent form.
Arm/Group | Nemolizumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 10
  White | 7
  Other: Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Nemolizumab Serum Concentrations at Week 1-2
Description: Serum concentrations of Nemolizumab were analyzed using validated enzyme linked immunosorbent assay (ELISA).
Time Frame: At week 1-2
Population: The pharmacokinetic (PK) population included all participants in the Safety population who provided at least 1 post-baseline evaluable drug concentration value. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Nemolizumab
Number analyzed (Participants) | 17
nanogram per milliliter (ng/mL) | 6478.8 (2393.11)

2. Primary Outcome: Nemolizumab Serum Concentrations at Week 4
Description: Serum concentrations of Nemolizumab were analyzed using validated enzyme linked immunosorbent assay (ELISA).
Time Frame: At week 4
Population: PK population included all participants in the Safety population who provided at least 1 post-baseline evaluable drug concentration value. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 17
ng/mL | 2935.3 (1029.41)

3. Primary Outcome: Nemolizumab Serum Concentrations at Week 8
Description: Serum concentrations of Nemolizumab were analyzed using validated enzyme linked immunosorbent assay (ELISA).
Time Frame: At week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 15
ng/mL | 3292.3 (2017.83)

4. Primary Outcome: Nemolizumab Serum Concentrations at Week 12
Description: Serum concentrations of Nemolizumab were analyzed using validated enzyme linked immunosorbent assay (ELISA).
Time Frame: At week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 14
ng/mL | 3221.6 (1781.15)

5. Primary Outcome: Nemolizumab Serum Concentrations at Week 16
Description: Serum concentrations of Nemolizumab were analyzed using validated enzyme linked immunosorbent assay (ELISA).
Time Frame: At week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 13
ng/mL | 3010.0 (1131.81)

6. Primary Outcome: Nemolizumab Serum Concentrations at Week 24
Description: Serum concentrations of Nemolizumab were analyzed using validated enzyme linked immunosorbent assay (ELISA).
Time Frame: At week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 8
ng/mL | 473.9 (333.72)

7. Primary Outcome: Apparent Clearance After Extravascular Administration (Cl/F) of Nemolizumab
Description: CL/F is apparent clearance of the drug from the serum, calculated as the drug dose divided area under the curve from time 0 extrapolated to infinite time [AUC (0-inf)].
Time Frame: Baseline to week 24
Population: PK population included all participants in the Safety population who provided at least 1 post-baseline evaluable drug concentration value.
Measure: Mean (Standard Deviation); unit: liter/day (L/day)
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
liter/day (L/day) | 0.325 (0.153)

8. Primary Outcome: Apparent Volume of Distribution After Extravascular Administration (Vd/F) of Nemolizumab
Description: Vd/F was calculated as dose divided by lambda_z *AUC(0-inf).
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
liter | 7.15 (2.24)

9. Primary Outcome: Population Lag Time (Tlag)
Description: Lag time is defined as the time taken for a drug to appear in the systemic circulation following administration. The population Tlag value was estimated for the overall population and was reported in this endpoint.
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
hours | 1.0728 (0)

10. Primary Outcome: First Order Constant of Absorption (ka)
Description: PK of Nemolizumab was evaluated in participants using Ka using PK samples collected on Weeks 1-2, 4, 8, 12, 16 and 24. Ka was evaluated by population PK (popPK) methods and mean and standard from the model has been tabulated.
Time Frame: Baseline to week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 1/day
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
1/day | 0.402 (0.145)

11. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Nemolizumab
Description: Cmax was obtained from serum concentration time curve.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 12
ng/mL | 5975.5 (2175.2)

12. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of Nemolizumab
Description: Time to reach maximum observed serum concentration (Tmax) for Nemolizumab was derived from serum concentrations versus time data.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nemolizumab
Number analyzed (Participants) | 12
days | 5.862 (1.669)

13. Primary Outcome: Trough Serum Concentration (Ctrough) of Nemolizumab at Week 4
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: At week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 17
ng/mL | 3271.859 (1268.612)

14. Primary Outcome: Trough Serum Concentration (Ctrough) of Nemolizumab at Week 8
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: At week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 14
ng/mL | 3056.496 (1367.884)

15. Primary Outcome: Trough Serum Concentration (Ctrough) of Nemolizumab at Week 12
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: At week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 14
ng/mL | 2886.796 (1441.998)

16. Primary Outcome: Trough Serum Concentration (Ctrough) of Nemolizumab at Week 16
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: At week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 12
ng/mL | 2981.792 (1166.871)

17. Primary Outcome: Area Under the Serum Concentration-Time Curve From Zero to 4 Week Post-dose (AUC0-4w)
Description: Area under the drug concentration-time curve from 0 to 4 week post dosing for Nemolizumab. AUC(0-4w) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose through 4 weeks post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram*day per milliliter (ng*day/mL)
Arm/Group | Nemolizumab
Number analyzed (Participants) | 17
nanogram*day per milliliter (ng*day/mL) | 144046.235 (50800.805)

18. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to 8 Week Post-dose (AUC0-8w)
Description: Area under the drug concentration-time curve from 0 to 8 week post dosing for Nemolizumab. AUC(0-8w) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose through 8 weeks post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 14
ng*day/mL | 284397.143 (97105.285)

19. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to 12 Week Post-dose (AUC0-12w)
Description: Area under the drug concentration-time curve from 0 to 12 week post dosing for Nemolizumab. AUC(0-12w) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose through 12 week post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 14
ng*day/mL | 411707.857 (142851.408)

20. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to 16 Week Post-dose (AUC0-16w)
Description: Area under the drug concentration-time curve from 0 to 16 week post dosing for Nemolizumab. AUC(0-16w) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose through 16 weeks post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 12
ng*day/mL | 549489.167 (184483.765)

21. Primary Outcome: Apparent Terminal Half-life (t1/2)
Description: Apparent Terminal Half-life (t1/2) is the time required for a given drug concentration in the serum to decrease by 50%.
Time Frame: Baseline to week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
day | 16.666 (4.115)

22. Primary Outcome: Number of Participants With Treatment-Related Positive Anti-Drug Antibodies (ADA) in Serum at Week 4
Description: Antidrug antibodies were determined using a validated enzyme-linked immunosorbent assay (ELISA) assay. Number of participants with positive ADA in Serum were reported.
Time Frame: At week 4
Population: The Safety population included all participants in ITT population who were administered at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Participants | 1

23. Primary Outcome: Number of Participants With Neutralizing Antibodies
Description: The number of participants with neutralizing antibodies response at time of baseline up to week 24 has been presented. Neutralizing antibodies response assay result have been only presented for participants with positive anti-drug antibody assay.
Time Frame: Baseline up to Week 24
Population: The safety population included all participants in the ITT who were administered at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Participants | 0

24. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Adverse Event of Special Interests (AESI) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAE was defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs. An AESI is a noteworthy event for study drug that should be monitored closely and reported immediately. The following AEs will be considered AESIs: Anaphylactic reactions, Acute allergic reactions requiring treatment, Severe injection site reaction, Newly-diagnosed asthma or worsening of asthma, Peripheral edema: limbs, bilateral and Facial edema.
Time Frame: Baseline through week 24
Population: The Safety population included all participants in the ITT who were administered at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Participants
  TEAEs | 6
  TE-AESIs | 2
  SAEs | 2

25. Primary Outcome: Number of Participants With Asthma Control Test (ACT) Score Less Than or Equal to (=<) 19 at Week 1-2
Description: The ACT is a participant-completed assessment consisting of 5 questions health survey for measuring asthma control. Each question is answered with a score in a range of 1 to 5 and lower score represents the more severe condition. The scale range for Question 1 is "all the time" (1) to "none of the time" (5); Question 2 range: "more than once a day" (1) to "not at all" (5); Question 3 range: "4 or more nights a week" (1) to "not at all" (5); Question 4 range: "3 or more times per day" (1) to "not at all" (5); Question 5 range: "not controlled at all" (1) to "completely controlled" (5). A total ACT score is obtained as the sum of the 5 individual question scores that is from 5 to 25, where Higher scores mean that asthma is more controlled.
Time Frame: At week 1-2
Population: Safety population included all participants in the ITT set who were administered at least 1 dose of study medication. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 10
Participants | 0

26. Primary Outcome: Number of Participants With Asthma Control Test (ACT) Score Less Than or Equal to (=<) 19 at Week 4
Description: as for outcome 25
Time Frame: At week 4
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 8
Participants | 0

27. Primary Outcome: Number of Participants With Asthma Control Test (ACT) Score Less Than or Equal to (=<) 19 at Week 8
Description: as for outcome 25
Time Frame: At week 8
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 7
Participants | 0

28. Primary Outcome: Number of Participants With Asthma Control Test (ACT) Score Less Than or Equal to (=<) 19 at Week 12
Description: as for outcome 25
Time Frame: At week 12
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 7
Participants | 1

29. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination (PE) Findings
Description: A complete PE included assessments of the head, ears, eyes, nose, throat, neck (including thyroid), skin/integumentary system, cardiovascular system, respiratory system, gastrointestinal system, musculoskeletal system, lymph nodes, and nervous system. Clinical significance was determined by the investigator.
Time Frame: Baseline up to Week 24
Population: Safety population included all participants in the ITT set who were administered at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Participants | 2

30. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Values
Description: Laboratory investigation included hematology, biochemistry, and urinalysis. Clinical significance was determined by the investigator. The number of participants with clinically significant abnormalities in laboratory parameters were reported.
Time Frame: Baseline up to Week 24
Population: Safety population included all participants in the ITT set who were administered at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Participants
  Hematology | 6
  Biochemistry | 5
  Urinalyses | 0

31. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Findings at Week 16
Description: The ECG recordings were obtained after 10 minutes of rest in a semi-supine position. Number of participants with clinically significant change from baseline in ECG findings were reported. Clinically significance was decided by investigator.
Time Frame: At week 16
Population: Safety population included all participants in the ITT set who were administered at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Participants | 0

32. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs included pulse rate, systolic and diastolic blood pressure (after the participant had been sitting for at least 5 minutes), and body temperature. Clinically significance was decided by investigator..
Time Frame: Baseline up to Week 24
Population: Safety population included all participants in the ITT set who were administered at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Participants | 5

33. Primary Outcome: Number of Participants With Abnormal Peak Expiratory Flow (PEF) <80% of Predicted Value at Week 1-2
Description: PEF was the maximum speed of expiration measured using spirometer. A participant took rest just before the measurement. At each time of measurement, a participant expired for at least 6 seconds wherever possible. At each time of measurement, at least 3 readings were obtained, and three readings which were obtained in an appropriate manner were stored. PEF <80% of predictive value is considered as abnormal.
Time Frame: At week 1-2
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 10
Participants | 1

34. Primary Outcome: Number of Participants With Abnormal Peak Expiratory Flow (PEF) <80% Predicted Value at Week 4
Description: as for outcome 33
Time Frame: At week 4
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 8
Participants | 1

35. Secondary Outcome: Non-Compartmental Analysis: Area Under the Serum Concentration-time Curve From Time Zero to 4 Weeks Post-dose AUC(0-4w)
Description: as for outcome 17
Time Frame: Pre-dose through 4 weeks post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 17
ng*day/mL | 122286.736 (44081.623)

36. Secondary Outcome: Non-Compartmental Analysis: Area Under the Serum Concentration-Time Curve From Time Zero to 8 Week Post-dose (AUC0-8w)
Description: as for outcome 18
Time Frame: Pre-dose through 8 weeks post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 13
ng*day/mL | 233258.841 (80113.408)

37. Secondary Outcome: Non-Compartmental Analysis: Area Under the Serum Concentration-Time Curve From Time Zero to 12 Week Post-dose (AUC0-12w)
Description: as for outcome 19
Time Frame: Pre-dose through 12 week post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 13
ng*day/mL | 332928.434 (121739.832)

38. Secondary Outcome: Non-Compartmental Analysis: Area Under the Serum Concentration-Time Curve From Time Zero to 16 Week Post-dose (AUC0-16w)
Description: as for outcome 20
Time Frame: Pre-dose through 16 weeks post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Nemolizumab
Number analyzed (Participants) | 12
ng*day/mL | 372858.017 (149908.126)

39. Secondary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 16
Description: EASI assesses severity and extent of atopic dermatitis (AD) signs through a composite score of erythema, induration/population, excoriation, and lichenification. Each characteristic was assessed for severity on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs. The total EASI score range from 0 to 72 with higher scores representing greater severity of AD.
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants who signed informed consent form. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
units on a scale | -15.994 (9.9413)

40. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 16
Description: EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. Each characteristic was assessed for severity on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs. The EASI score can range from 0 to 72 with higher scores representing greater severity of AD.
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Percent change | -66.52 (32.461)

41. Secondary Outcome: Number of Participants Who Achieved Investigator's Global Assessment (IGA) Success (Defined as IGA 0 [Clear] or 1 [Almost Clear]) From Baseline to Week 16
Description: IGA is a 5-point scale used by the investigator or trained designee to evaluate the global severity of AD. Ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), where higher score indicated higher severity. IGA success is defined as participants with 0 (clear) or 1 (almost clear) and at least 2 -grade improvement from baseline. Number of Participants who achieved Investigator's Global Assessment (IGA) Success from baseline to week 16 were reported.
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants who signed informed consent form.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab
Number analyzed (Participants) | 20
Participants | 7

42. Secondary Outcome: Change From Baseline in the Percentage of Body Surface Area (BSA) Involvement by Atopic Dermatitis (AD) at Each Visit up to Week 24
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and reported as a percentage of all major body sections combined. The reported percentage of BSA was combined percentage of all major body sections.
Time Frame: Baseline, Week 1-2, 4, 8, 12, 14, 16 and 24
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Percentage of BSA
  Week 1 to 2 | -1.9 (6.33)
  Week 4 | -7.1 (15.90)
  Week 8 | -11.2 (15.48)
  Week 12 | -17.2 (17.94)
  Week 16 | -19.9 (17.04)
  Week 24 | -14.7 (17.88)

43. Secondary Outcome: Absolute Change From Baseline in Weekly Average of Peak Pruritus Numeric Rating Scale (NRS) Score at Week 16
Description: Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity.
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
score on a scale | -3.122 (2.8216)

44. Secondary Outcome: Percent Change From Baseline in Weekly Average of Peak Pruritus Numeric Rating Scale (NRS) Score at Week 16
Description: as for outcome 43
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Percent of change
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Percent of change | -43.21 (36.970)

45. Secondary Outcome: Absolute Change From Baseline in Weekly Average of Average Pruritus Numeric Rating Scale (NRS) Score at Week 16
Description: as for outcome 43
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
score on a scale | -2.610 (2.6148)

46. Secondary Outcome: Percent Change From Baseline in Weekly Average of Average Pruritus Numeric Rating Scale (NRS) Score at Week 16
Description: as for outcome 43
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Percent change | -40.85 (37.293)

47. Secondary Outcome: Absolute Change From Baseline in Weekly Average Sleep Disturbance Numeric Rating Scale (NRS) Score at Week 16
Description: The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants were asked the following questions in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Higher scores indicate worse outcome.
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
score on a scale | -3.050 (3.2367)

48. Secondary Outcome: Percent Change From Baseline in Weekly Average Sleep Disturbance Numeric Rating Scale (NRS) Score at Week 16
Description: as for outcome 47
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Nemolizumab
Number analyzed (Participants) | 18
Percent change | -53.51 (47.782)

49. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Week 16
Description: Scoring Atopic Dermatitis (SCORAD) is a validated measure commonly used to assess the severity and the extent of AD signs and symptoms. SCORAD is a clinical tool for assessing the severity and the extent of AD signs and symptoms. Extent and intensity of six types of basic lesions (erythema/darkening, edema/papule, oozing/crusting, excoriation, lichenification/prurigo and dryness) and symptoms (itching and loss of sleep) were assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Baseline, Week 16
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Nemolizumab
Number analyzed (Participants) | 20
Percent change | -50.08 (26.925)

50. Secondary Outcome: Number of Topical Atopic Dermatitis Medication-Free Days Through Week 24
Description: Number of topical AD medication-free days through Week 16 was calculated as the number of days that a participant used neither topical corticosteroid (TCS)/ topical calcineurin inhibitors (TCI) nor system rescue therapy divided by the study days.
Time Frame: Baseline through Week 24
Population: ITT population included all enrolled participants who signed informed consent form. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here "Number analyzed" signifies those participants who were evaluable for this outcome measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nemolizumab
Number analyzed (Participants) | 20
Days
  Baseline to Week 1-2: number analyzed (Participants) | 19
  Baseline to Week 1-2 | 3.5 (2.25)
  Week 1-2 to Week 4: number analyzed (Participants) | 19
  Week 1-2 to Week 4 | 7.5 (4.87)
  Week 4 to Week 8: number analyzed (Participants) | 18
  Week 4 to Week 8 | 12.1 (7.20)
  Week 8 to Week 12: number analyzed (Participants) | 15
  Week 8 to Week 12 | 9.7 (5.96)
  Week 12 to Week 16: number analyzed (Participants) | 15
  Week 12 to Week 16 | 10.7 (5.82)
  Week 16 to Week 24: number analyzed (Participants) | 14
  Week 16 to Week 24 | 23.4 (11.88)

51. Secondary Outcome: Dermatology Life Quality Index (DLQI) For Participants > 16 Years of Age at Baseline and Week 16
Description: The DLQI is a validated 10-item questionnaire covering domains including symptoms/feelings, daily activities, leisure, work/school, personal relationships, and treatment. The participants were rate each question ranging from 0 (not at all) to 3 (very much) and overall score ranges from 0 to 30. A higher total score indicates a poorer quality of life (QoL).
Time Frame: Baseline, Week 16
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nemolizumab
Number analyzed (Participants) | 5
score on a scale
  Baseline | 11.8 (3.11)
  Week 16: number analyzed (Participants) | 4
  Week 16 | 3.0 (2.58)

52. Secondary Outcome: Children's Dermatology Life Quality Index (cDLQI) For Participants 12-16 Years of Age at Baseline and Week 16
Description: as for outcome 51
Time Frame: Baseline, Week 16
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nemolizumab
Number analyzed (Participants) | 13
score on a scale
  Baseline | 10.6 (5.42)
  Week 16: number analyzed (Participants) | 10
  Week 16 | 6.2 (5.29)

ADVERSE EVENTS:
Time Frame: Baseline through Week 24
Description: Safety population included all participants in the ITT set who were administered at least 1 dose of study medication.
Arm/Group | Nemolizumab
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemolizumab (N=18)
Oedema peripheral (General disorders) | 1 (1)
Eczema infected (Infections and infestations) | 1 (1)
Staphylococcus skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab (N=18)
Oedema peripheral (General disorders) | 1
Fatigue (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03921411/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03921411/SAP_001.pdf